CLINICAL TRIAL: NCT00346814
Title: Antiangiogenic Therapy With Bevacizumab in Retinopathy of Prematurity. Structural Outcome
Status: Recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Asociación para Evitar la Ceguera en México (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: APEC-001
Record Dates: First submitted 2006-06-29; First posted 2006-06-30 (Estimated); Last update posted 2024-07-31 (Actual); Status verified 2024-07

CONDITIONS: Retinopathy of Prematurity
Keywords: Retinopathy of prematurity; antiangiogenic therapy
MeSH Terms: conditions — Retinopathy of Prematurity | interventions — Intravitreal Injections

INTERVENTIONS:
Drug: intravitreal injection

SUMMARY:
Purpose:Retinopathy of prematurity (ROP) continues tobe a major cause of blindness in children. Although ablation of the retina with laser or cryotherapy reduces the incidence of blindness by suppressing the neovascular phase of ROP the visual outcomes after treatment are often poor. Vascular endothelial growth factor(VEGF) has an important role in the pathogenesis of ROP and inhibition of VEGF expression in the neovascular phase might prevent destructive neovascularization in ROP. The aim of this study is to determine the safety and efficacy of intravitreal bevacizumab in the treatment of retinopathy of prematurity

ELIGIBILITY:
Inclusion Criteria:

* Retinopathy of prematurity stages III, IV and V in which we can not treat with laser o cryotherAPY

Exclusion Criteria:

* PATIENTS THAT COULD BE TREATED WITH CRYOTHERAPY OR LASER

Ages: 1 Month to 12 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Dates: Start 2007-07 (Actual); Primary Completion 2007-07 (Actual); Study Completion 2024-11 (Estimated)

PRIMARY OUTCOMES:
Clinical appearance

CONTACTS AND LOCATIONS:
Overall Officials: Maria Martínez-Castellanos, MD, Principal Investigator — Asociación para Evitar la Ceguera en México
Locations (1):
- Asociación para Evitar la Ceguera en México Hospital "Luis Sanchez Bulnes", Mexico City, Mexico DF, Mexico